CLINICAL TRIAL: NCT01794780
Title: A 1-year Multi-center, Prospective, Cohort Study in Patients With Chronic Obstructive Pulmonary Disease Treated With Long-acting Bronchodilator
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CQAB149BCN01
Record Dates: First submitted 2013-02-15; First posted 2013-02-20 (Estimated); Results first posted 2019-09-26 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-08

CONDITIONS: COPD
Keywords: COPD; Chronic obstructive pulmonary disease (COPD),; Chronic obstructive lung disease (COLD),; Chronic obstructive airway disease (COAD),; Cronchitis,; Emphysema
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema | interventions — Fluticasone; Formoterol Fumarate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Indacaterol (Experimental): LABA: Indacaterol, once a day, 150μg each time
  Interventions: Drug: LABA based treatment: indacaterol
- Tiotropium Bromide (Experimental): LAMA: Tiotropium Bromide, once a day, 18 μg
  Interventions: Drug: LAMA based treatment: tiotropium
- Salmeterol/Fluticasone (Experimental): LABA/ICS: Salmeterol/Fluticasone, twice a day, 50/250 μg, 50/500 μg
  Interventions: Drug: LABA/ICS based treatment: salmeterol/fluticasone
- Budesonide/ formoterol (Experimental): Budesonide/formoterol, twice daily, two suction each time, 160/4.5 μg
  Interventions: Drug: LABA/ICS based treatment: budesonide/formoterol
- Indacaterol +Tiotropium (Experimental): Indacaterol, once a day, 150μg each time +Tiotropium Bromide, once a day, 18 μg
  Interventions: Drug: LABA based treatment: indacaterol; Drug: LAMA based treatment: tiotropium
- LABA/ICS (Or budesonide/ formoterol)+ Tiotropium (Experimental): Salmeterol / fluticasone Or budesonide / formoterol
  Interventions: Drug: LAMA based treatment: tiotropium; Drug: LABA/ICS based treatment: salmeterol/fluticasone; Drug: LABA/ICS based treatment: budesonide/formoterol
- Oral theophylline (Experimental)
  Interventions: Drug: theophylline based treatment
- Other treatment (Experimental): non-long-acting bronchodilators for COPD treatment, such treatments were classified as "other treatments"
  Interventions: Drug: Other treatment

INTERVENTIONS:
Drug: LABA based treatment: indacaterol — LABA based treatment: indacaterol
  Arms: Indacaterol; Indacaterol +Tiotropium
Drug: LAMA based treatment: tiotropium — LAMA based treatment: tiotropium
  Arms: Indacaterol +Tiotropium; LABA/ICS (Or budesonide/ formoterol)+ Tiotropium; Tiotropium Bromide
Drug: LABA/ICS based treatment: salmeterol/fluticasone — LABA/ICS based treatment: salmeterol/fluticasone
  Arms: LABA/ICS (Or budesonide/ formoterol)+ Tiotropium; Salmeterol/Fluticasone
Drug: LABA/ICS based treatment: budesonide/formoterol — LABA/ICS based treatment: budesonide/formoterol
  Arms: Budesonide/ formoterol; LABA/ICS (Or budesonide/ formoterol)+ Tiotropium
Drug: theophylline based treatment — theophylline based treatment
  Arms: Oral theophylline
Drug: Other treatment — non-long-acting bronchodilators for COPD treatment, such treatments were classified as "other treatments"
  Arms: Other treatment

SUMMARY:
This multi-center study is designed to describe natural history of disease, treatment and health care products in physician-diagnosed COPD patients who require adding daily maintenance therapy in real world.

The study planned to enroll 550 patients in Indacaterol group and 9450 patients in non- Indacaterol group, a total of 10,000 patients. Enrollment was stopped at 2253 patients due to low recruitment in indacaterol group. Finally a total of 2229 patients were analyzed in full analysis set.

A total of 2253 patients entered into the database, of which 24 patients were exclude during the data review meetings, because they did not met the inclusion/exclusion criteria. Hence a total of 2229 patients enrolled successfully.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent
* Physician-diagnosis of COPD
* COPD patients requiring long-acting bronchodilator treatment
* Patients with spirometry available at baseline

Exclusion Criteria:

* Patients who have a diagnosis of asthma.
* Patients who had been hospitalized for a COPD exacerbation in the 4 weeks prior to Visit 1.
* Current clinical diagnosis of other chronic respiratory illnesses
* Concurrent participation in a clinical trial or use of an investigational drug.
* Active malignancy or history of malignancy of any organ system
* Pregnant or nursing (lactating) women
* Women of child-bearing potential with no contraception Other protocol-defined inclusion/exclusion criteria may apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2229 (Actual)
Dates: Start 2013-02-05 (Actual); Primary Completion 2015-05-25 (Actual); Study Completion 2015-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- China (2):
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Zhengzhou

REFERENCES:
- [Derived] Han J, Dai L, Zhong N, Young D. Breathlessness or health status in chronic obstructive pulmonary disease: the impact of different definitions. COPD. 2015 Apr;12(2):115-25. doi: 10.3109/15412555.2014.974741. Epub 2014 Dec 4. PMID 25474373

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 2253 patients entered into the database, of which 24 patients were exclude during the data review meetings, because they did not met the inclusion/exclusion criteria. Hence a total of 2229 patients enrolled successfully.
Groups:
- Oral Theophylline: Oral theophylline
Period: Overall Study
Arm/Group | Indacaterol | Tiotropium Bromide | Salmeterol/Fluticasone | Budesonide/ Formoterol | Indacaterol +Tiotropium | LABA/ICS (Or Budesonide/ Formoterol)+ Tiotropium | Oral Theophylline | Other Treatment
Started | 32 | 276 | 813 | 283 | 9 | 632 | 154 | 30
Completed | 15 | 180 | 571 | 200 | 6 | 452 | 112 | 21
Not Completed | 17 | 96 | 242 | 83 | 3 | 180 | 42 | 9
Not completed — Adverse Event | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 2 | 14 | 1 | 0 | 9 | 4 | 0
Not completed — Lost to Follow-up | 10 | 64 | 165 | 53 | 2 | 99 | 30 | 5
Not completed — Withdrew informed consent | 7 | 17 | 36 | 9 | 0 | 48 | 4 | 3
Not completed — Other | 0 | 12 | 25 | 20 | 1 | 24 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Indacaterol | Tiotropium Bromide | Salmeterol/Fluticasone | Budesonide/ Formoterol | Indacaterol +Tiotropium | LABA/ICS (Or Budesonide/ Formoterol)+ Tiotropium | Oral Theophylline | Other Treatment | Total
Number analyzed (Participants) | 32 | 276 | 813 | 283 | 9 | 632 | 154 | 30 | 2229
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.12 (9.238) | 68.93 (9.145) | 67.00 (9.353) | 67.02 (9.858) | 69.49 (8.873) | 67.74 (9.427) | 67.86 (9.652) | 66.14 (10.205) | 67.50 (9.453)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 52 | 154 | 49 | 1 | 81 | 35 | 5 | 378
  Male | 31 | 224 | 659 | 234 | 8 | 551 | 119 | 25 | 1851

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1)
Description: Forced expiratory volume in 1 second (FEV1) is the amount of air that can be exhaled in one second. A positive change from baseline in FEV1 indicates improvement in lung function. Pulmonary function tests were performed at study visits including FEV1, and Force Vital Capacity (FVC). These were performed 30 minutes before treatment and not more than 2 hours in advance after stopping the Long-acting bronchodilators eight hours before visits. In order to reduce the variation between each test, the same instrument was used in the whole research process if condition allowed.
Time Frame: Baseline,3 months
Population: FAS: Two Arms/Groups were grouped together in the analysis as some of the analysis required to combine the results. Per protocol it was not the intent to compare the results between different standard of care (LABA/ICS). Efficacy data were not collected separately for the "Salmeterol / fluticasone" and "budesonide / formoterol" Arms/Groups,"
Measure: Mean (Standard Deviation); unit: Liters
Groups:
- Tiotropium: LAMA: Tiotropium Bromide, once a day, 18 μg
- LABA/ICS: Salmeterol / fluticasone Or budesonide / formoterol
- Indacaterol + Tiotropium: Indacaterol, once a day, 150μg each time +Tiotropium Bromide, once a day, 18 μg
- LABA/ICS + Tiotropium: (Salmeterol / fluticasone Or budesonide / formoterol) + tiotropium
Arm/Group | Indacaterol | Tiotropium | LABA/ICS | Indacaterol + Tiotropium | LABA/ICS + Tiotropium | Oral Theophylline
Number analyzed (Participants) | 22 | 154 | 702 | 6 | 404 | 104
Liters | -0.042 (0.1742) | 0.006 (0.2537) | 0.033 (0.3790) | 0.022 (0.1157) | 0.011 (0.2417) | 0.012 (0.3405)

2. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1)
Description: as for outcome 1
Time Frame: Baseline,12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Indacaterol | Tiotropium Bromide | LABA/ICS | Indacaterol +Tiotropium | LABA/ICS + Tiotropium | Oral Theophylline
Number analyzed (Participants) | 10 | 129 | 597 | 3 | 317 | 87
Liters | 0.056 (0.2137) | -0.036 (0.2395) | 0.056 (0.4335) | 0.030 (0.0854) | -0.028 (0.2258) | 0.046 (0.3654)

3. Secondary Outcome: COPD Exacerbation
Description: Number of COPD exacerbations evaluated over 12 months. COPD exacerbation is defined as a new onset or worsening of at least 1 respiratory major symptoms (e.g. dyspnea, cough, sputum volume or sputum purulence) for at least 3 consecutive days, which results in recorded treatment change (antibiotics/steroids/oxygen therapy) OR recorded COPD related hospitalization/Emergency visit. COPD exacerbation is not considered as adverse event, and should only be recorded in COPD e-CRF.
Time Frame: Baseline,12 months
Population: FAS: Two Arms/Groups were grouped together in the analysis as some of the analysis required to combine the results. Per protocol it was not the intent to compare the results between different standard of care (LABA/ICS)
Measure: Mean (Standard Deviation); unit: COPD Exacerbations/year
Arm/Group | Indacaterol | Tiotropium Bromide | Salmeterol/Fluticasone | Budesonide/ Formoterol | LABA/ICS | Indacaterol +Tiotropium | LABA/ICS + Tiotropium | Oral Theophylline
Number analyzed (Participants) | 32 | 276 | 813 | 283 | 1096 | 9 | 632 | 154
COPD Exacerbations/year | 1.1 (3.53) | 0.5 (1.89) | 1.1 (7.74) | 0.4 (1.89) | 0.9 (6.72) | 4.1 (5.46) | 0.8 (3.47) | 1.0 (3.57)

4. Secondary Outcome: Change in Health Status Questionnaire MMRC
Description: The mMRC scale is scored from 0 (less severe) to 4 (severe). 0 Not troubled with breathlessness except with strenuous exercise; 1 Troubled by shortness of breath when hurrying on the level or walking up a slight hill; 2 Walks slower than people of the same age on the level because of breathlessness or has to stop for breath when walking at own pace on the level; 3 Stops for breath after walking about 100 yards or after a few minutes on the level; 4 Too breathless to leave the house or breathless when dressing or undressing. The modified Medical Research Council (mMRC) Dyspnea Scale , is a five-item instrument (part of the Borg scale) to assess a patient's degree of breathlessness in relation to physical activity. Participants will be required to read a brief description of an activity and then select a statement that best describes their experience with dyspnea at Visit 101. The mMRC was assessed by the investigators at the scheduled visits.
Time Frame: Baseline,3,6,9,12 months
Population: FAS: Two Arms/Groups were grouped together in the analysis as some of the analysis required to combine the results. Per protocol it was not the intent to compare the results between different standard of care (LABA/ICS).Efficacy data were not collected separately for the "Salmeterol / fluticasone" and "budesonide / formoterol" Arms/Groups,"
Measure: Number; unit: Number of participants
Arm/Group | Indacaterol | Tiotropium Bromide | LABA/ICS | Indacaterol +Tiotropium | LABA/ICS + Tiotropium | Oral Theophylline
Number analyzed (Participants) | 32 | 276 | 1096 | 9 | 632 | 154
Number of participants
  Baseline scale item 0 | 4 | 40 | 161 | 1 | 63 | 31
  Baseline scale item 1 | 11 | 114 | 435 | 4 | 226 | 66
  Baseline scale item 2 | 14 | 83 | 327 | 1 | 211 | 34
  Baseline scale item 3 | 3 | 36 | 154 | 3 | 110 | 19
  Baseline scale item 4 | 0 | 3 | 19 | 0 | 22 | 4
  3 month Scale item 0: number analyzed (Participants) | 20 | 167 | 741 | 7 | 411 | 110
  3 month Scale item 0 | 3 | 24 | 101 | 0 | 54 | 20
  3 month Scale item 1: number analyzed (Participants) | 20 | 167 | 741 | 7 | 411 | 110
  3 month Scale item 1 | 9 | 69 | 364 | 4 | 157 | 52
  3 month Scale item 2: number analyzed (Participants) | 20 | 167 | 741 | 7 | 411 | 110
  3 month Scale item 2 | 7 | 54 | 203 | 3 | 133 | 26
  3 month Scale item 3: number analyzed (Participants) | 20 | 167 | 741 | 7 | 411 | 110
  3 month Scale item 3 | 1 | 18 | 67 | 0 | 58 | 11
  3 month Scale item 4: number analyzed (Participants) | 20 | 167 | 741 | 7 | 411 | 110
  3 month Scale item 4 | 0 | 2 | 6 | 0 | 9 | 1
  6 month Scale item 0: number analyzed (Participants) | 16 | 141 | 583 | 6 | 346 | 82
  6 month Scale item 0 | 2 | 23 | 96 | 0 | 37 | 15
  6 month Scale item 1: number analyzed (Participants) | 16 | 141 | 583 | 6 | 346 | 82
  6 month Scale item 1 | 5 | 57 | 290 | 1 | 149 | 43
  6 month Scale item 2: number analyzed (Participants) | 16 | 141 | 583 | 6 | 346 | 82
  6 month Scale item 2 | 8 | 45 | 138 | 4 | 105 | 20
  6 month Scale item 3: number analyzed (Participants) | 16 | 141 | 583 | 6 | 346 | 82
  6 month Scale item 3 | 1 | 13 | 54 | 1 | 44 | 4
  6 month Scale item 4: number analyzed (Participants) | 16 | 141 | 583 | 6 | 346 | 82
  6 month Scale item 4 | 0 | 3 | 5 | 0 | 11 | 0
  9 month Scale item 0: number analyzed (Participants) | 13 | 121 | 549 | 3 | 321 | 85
  9 month Scale item 0 | 3 | 24 | 116 | 0 | 45 | 20
  9 month Scale item 1: number analyzed (Participants) | 13 | 121 | 549 | 3 | 321 | 85
  9 month Scale item 1 | 5 | 52 | 256 | 1 | 127 | 40
  9 month Scale item 2: number analyzed (Participants) | 13 | 121 | 549 | 3 | 321 | 85
  9 month Scale item 2 | 4 | 30 | 131 | 2 | 99 | 19
  9 month Scale item 3: number analyzed (Participants) | 13 | 121 | 549 | 3 | 321 | 85
  9 month Scale item 3 | 1 | 14 | 42 | 0 | 41 | 5
  9 month Scale item 4: number analyzed (Participants) | 13 | 121 | 549 | 3 | 321 | 85
  9 month Scale item 4 | 0 | 1 | 4 | 0 | 9 | 1
  12 month Scale item 0: number analyzed (Participants) | 10 | 131 | 602 | 3 | 328 | 89
  12 month Scale item 0 | 1 | 24 | 150 | 0 | 47 | 20
  12 month Scale item 1: number analyzed (Participants) | 10 | 131 | 602 | 3 | 328 | 89
  12 month Scale item 1 | 5 | 61 | 275 | 2 | 138 | 52
  12 month Scale item 2: number analyzed (Participants) | 10 | 131 | 602 | 3 | 328 | 89
  12 month Scale item 2 | 2 | 33 | 127 | 1 | 102 | 12
  12 month Scale item 3: number analyzed (Participants) | 10 | 131 | 602 | 3 | 328 | 89
  12 month Scale item 3 | 2 | 10 | 41 | 0 | 32 | 4
  12 month Scale item 4: number analyzed (Participants) | 10 | 131 | 602 | 3 | 328 | 89
  12 month Scale item 4 | 0 | 3 | 9 | 0 | 9 | 1

5. Secondary Outcome: Change From Baseline in Questionnaire COPD Assessment Test (CAT) Score
Description: The COPD assessment test (CAT) is a short instrument scale used to quantify the symptom burden of COPD and will be used to assess the health status of patients in this study. It consists of eight items, each presented as a semantic 6-point differential scale, providing a total score out of 40. A higher score indicates a worse health status. Scores of 0 - 10, 11 - 20, 21 - 30 and 31 - 40 represent a mild, moderate, severe or very severe clinical impact of COPD upon the patient.
Time Frame: Baseline,3,6,9,12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Indacaterol | Tiotropium Bromide | LABA/ICS | Indacaterol +Tiotropium | LABA/ICS + Tiotropium | Oral Theophylline
Number analyzed (Participants) | 32 | 276 | 1096 | 9 | 632 | 154
Score on a scale
  3 Month: number analyzed (Participants) | 20 | 167 | 741 | 7 | 411 | 110
  3 Month | -1.9 (5.12) | -2.1 (5.58) | -2.3 (5.68) | -1.9 (2.67) | -1.8 (5.96) | -1.8 (4.07)
  6 Month: number analyzed (Participants) | 16 | 140 | 582 | 6 | 346 | 82
  6 Month | -1.9 (5.80) | -2.7 (5.78) | -2.7 (5.89) | -2.7 (5.01) | -2.2 (6.46) | -2.5 (5.65)
  9 Month: number analyzed (Participants) | 13 | 121 | 549 | 3 | 321 | 85
  9 Month | -4.4 (5.27) | -3.1 (6.02) | -3.5 (6.66) | -9.0 (2.65) | -3.1 (6.49) | -3.1 (6.27)
  12 Month: number analyzed (Participants) | 10 | 131 | 603 | 3 | 328 | 89
  12 Month | -5.1 (3.98) | -2.6 (6.74) | -4.1 (7.09) | -7.7 (0.58) | -3.7 (6.45) | -2.4 (7.25)

6. Secondary Outcome: Change From Baseline Questionnaire Transition Dyspnea Index (TDI) Score
Description: Transition Dyspnea Index (TDI) captures changes from baseline. The TDI score is based on three domains with each domain scored from -3 (major deterioration) to +3 (major improvement), to give an overall score of -9 to +9, a negative score indicating a deterioration from baseline. A TDI focal score of 1 is considered to be a clinically significant improvement from baseline. BDI/TDI was used to assess dyspnea from several aspects, caused by daily activities. These were evaluated by the investigators in the study at the scheduled study visits. The indices were to be evaluated by the same investigator.as far as possible.
Time Frame: Baseline,3,6,9,12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- LABA/ICS + Tiotropium: Salmeterol / fluticasone Or budesonide / formoterol) + tiotropium
Arm/Group | Indacaterol | Tiotropium Bromide | LABA/ICS | Indacaterol +Tiotropium | LABA/ICS + Tiotropium | Oral Theophylline
Number analyzed (Participants) | 32 | 276 | 1096 | 9 | 632 | 154
Units on a scale
  Baseline: number analyzed (Participants) | 32 | 271 | 1078 | 9 | 624 | 150
  Baseline | 6.7 (2.27) | 6.6 (2.66) | 6.7 (2.66) | 5.4 (2.24) | 6.2 (2.60) | 7.1 (2.81)
  3 Month: number analyzed (Participants) | 19 | 167 | 740 | 7 | 411 | 110
  3 Month | 1.4 (2.61) | 1.2 (2.43) | 1.3 (2.59) | 0.4 (2.07) | 1.1 (2.50) | 0.9 (2.57)
  6 Month: number analyzed (Participants) | 16 | 141 | 582 | 6 | 345 | 82
  6 Month | 0.0 (2.45) | 1.0 (2.67) | 1.4 (2.59) | -0.5 (2.26) | 0.9 (2.36) | 1.2 (2.03)
  9 Month: number analyzed (Participants) | 12 | 119 | 549 | 3 | 320 | 85
  9 Month | 0.7 (1.23) | 0.9 (2.48) | 1.6 (2.78) | 1.0 (1.73) | 0.9 (2.32) | 1.4 (2.68)
  12 Month: number analyzed (Participants) | 10 | 131 | 604 | 3 | 328 | 89
  12 Month | 0.3 (1.70) | 1.0 (2.91) | 1.7 (3.09) | 1.0 (1.73) | 1.0 (2.57) | 1.6 (2.44)

ADVERSE EVENTS:
Groups:
- Indacaterol: Indacaterol
- Tiotropium: Tiotropium
- Salemeterol/Fluticasone: Salemeterol/Fluticasone
- Budesonide/Formoterol: Budesonide/Formoterol
- Indacaterol + Tiotropium: Indacaterol + Tiotropium
- Salemeterol/Fluticasone(or Budesonide/Formoterol)+Tiotropium: Salemeterol/Fluticasone(or Budesonide/Formoterol)+Tiotropium
- Other: Other
Arm/Group | Indacaterol | Tiotropium | Salemeterol/Fluticasone | Budesonide/Formoterol | Indacaterol + Tiotropium | Salemeterol/Fluticasone(or Budesonide/Formoterol)+Tiotropium | Oral Theophylline | Other
Serious Adverse Events (participants affected / at risk) | 1/32 | 9/276 | 22/813 | 2/283 | 2/9 | 11/632 | 6/154 | 1/30
Other Adverse Events (participants affected / at risk) | 2/32 | 1/276 | 14/813 | 1/283 | 1/9 | 5/632 | 1/154 | 1/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol (N=32) | Tiotropium (N=276) | Salemeterol/Fluticasone (N=813) | Budesonide/Formoterol (N=283) | Indacaterol + Tiotropium (N=9) | Salemeterol/Fluticasone(or Budesonide/Formoterol)+Tiotropium (N=632) | Oral Theophylline (N=154) | Other (N=30)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malignant lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute left ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0
Atrioventricular block (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac disorder (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertensive heart disease (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Unstable angina (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Positional vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Goitre (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Death (General disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Multi-organ failure (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sudden cardiac death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sudden death (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Abdominal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infectious pneumonia (Infections and infestations) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0
Spontaneous pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol (N=32) | Tiotropium (N=276) | Salemeterol/Fluticasone (N=813) | Budesonide/Formoterol (N=283) | Indacaterol + Tiotropium (N=9) | Salemeterol/Fluticasone(or Budesonide/Formoterol)+Tiotropium (N=632) | Oral Theophylline (N=154) | Other (N=30)
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 14 | 1 | 0 | 4 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.